CLINICAL TRIAL: NCT05860049
Title: Adding Instrument Assisted Soft Tissue Mobilization to Core Stability Training in Chronic Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, RAGHDA MOHAMED HASSAN MAHMOUD, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003837
Record Dates: First submitted 2023-04-28; First posted 2023-05-16 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Core Stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional physiotherapy + Core stability (Active Comparator): They received conventional physical therapy and core stability for 4 weeks.
  Interventions: Other: Conventional physiotherapy; Other: Core stability
- Conventional physiotherapy + Core stability + Instrument assisted soft tissue mobilization (IASTM) (Experimental): They received conventional physical therapy, core stability, and IASTM technique for 4 weeks.
  Interventions: Other: Conventional physiotherapy; Other: Core stability; Device: Instrument assisted soft tissue mobilization

INTERVENTIONS:
Other: Conventional physiotherapy — All participants in both groups (A and B) received conventional physiotherapy program including infrared thermotherapy, transcutaneous electrical nerve stimulation, stretching exercises for for Upper Trapezius, Levator Scapulae, Sternocleidomastoid and Scalenes muscles, and active neck ROM exercises, 3 sessions per week, for 4 weeks.
Other: Core stability — All participants in both groups (A and B) received core stability exercises in the form of bridging exercise, bridging exercise on a ball, plank, and side plank 3 sessions per week, for 4 weeks.
Device: Instrument assisted soft tissue mobilization — Each participant in group (B) was seated in a comfortable position. The participant's forehead rested on his/her forearm on a table in front of him/her. A lubricant (Vaseline) was applied to the skin around the neck area prior to treatment, and the M2T blade (Figure 4) was cleaned with an alcohol pad. First, the M2T blade was used to find the exact areas of restriction in the RT upper trapezius. Then, the M2T blade was used at an angle of 45°, utilizing treatment planes 1, 2, and 3, to apply slow strokes along the muscle, without causing any discomfort or pain, from the muscle origin to its insertion for approximately 3 minutes. This procedure was repeated twice a week, for 4 weeks.
  Arms: Conventional physiotherapy + Core stability + Instrument assisted soft tissue mobilization (IASTM)

SUMMARY:
Purpose of the study was to investigate the effect of adding instrument assisted soft tissue mobilization to core stability training in treatment of chronic mechanical neck pain on pain level, cervical ROM, proprioception, muscle activity, H-reflex, and functions.

DETAILED DESCRIPTION:
Neck pain (NP) is a common musculoskeletal condition with a lifetime incidence rate between 22% and 70%.

Neck pain is commonly a recurrent condition with remissions and exacerbation that do not completely resolve. A history of previous injury to the neck (including whiplash, sports and work injuries etc.) increases the likelihood of chronic pain. As one ages, more chronic neck pain persists.

Mechanical neck pain is pain and/or stiffness in the neck or shoulder girdle region which was reproducible with neck movements.

Mechanical neck pain is the most common type found in neck-pain disorders. Studies have demonstrated altered behavior of the cervical muscles in mechanical neck-pain patients.

Mechanical neck pain produces mobility restriction, functional disability, decrease in muscle strength and decrease in health related quality of life.

Several treatment techniques and methods are used to rehabilitate pathologies of the cervical spine, including manual therapy, massage, stretching, soft-tissue techniques, and therapeutic exercise.

Manual therapy includes hands-on therapy techniques, such as soft tissue mobilization and massage techniques, as well as techniques using therapeutic equipment, such as stainless steel tools, that allow clinical therapists to identify and treat soft tissue dysfunctions.

Instrument-assisted soft tissue mobilization (IASTM) encompasses a broad range of techniques to treat soft tissue deficiencies. Tools used for IASTM produce micro-trauma to soft tissue for healing and restoring normal elasticity and function.

In recent years, Core stability training has become a popular fitness trend that has begun to be applied in rehabilitation programs and in sports medicine.

Core exercises have a positive effect on reducing lower back pain, improving upper extremities in breast cancer patients and lower extremities in patients with total hip and knee arthroplasty, as well as performance improvement for athletes. Core exercises are taken seriously in rehabilitation, medical care, and sports.

The core stability exercise program can be described as enhancing the ability to ensure a stable neutral spine position.

Statement of the problem Is there is effect of adding instrument assisted soft tissue mobilization to core stability in treatment of mechanical neck pain?

Purpose of the study:

Purpose of the study was to investigate effect of adding instrument assisted soft tissue mobilization to core stability in treatment of mechanical neck pain on pain level, cervical ROM, proprioception, muscle activity, H-reflex, and functions.

Significance of the study:

Study of Mohamed et al., (2020) investigated and compared the effects of instrument assisted soft tissue mobilization (IASTM) using m2t blade and trigger point release (TPR) in terms of neck lateral flexion and rotation range of motion on upper trapezius (UT) myofascial trigger points (MTrPs) in mechanical neck pain.

Both groups showed significant effects in improving range of motion. There was no significant difference in neck lateral flexion and rotation between the two groups.

The improvements in patients who received IASTM by M2t blade could be explained through loosening and removal of scar tissues and adhesions secondary to skin scraping which decreased soft tissue consistency and improved range of motion. It also induced vasodilation response and microvascular hemorrhage; so provided oxygen, nutrients and removed metabolic end products and inflammatory mediators which improved pain level and ppt.

Konstantinos et al., (2012) found that IASTM techniques combined with neuromuscular retraining exercises can significantly reduce pain and improve the corresponding function of patients with cervical pain compared to the application of the same exercises and a simple massage.

Rajalaxmi et al., (2020) analyzed the efficacy of multistep core stability exercise with and without conventional neck exercises in the treatment of chronic non-specific neck pain a Randomized Controlled Trial.

GROUP A received neck stability exercise and GROUP B received neck stability and core stability exercises. Both the groups received exercises for 45 min session per day for 6 days a week for 12 weeks. Pre and post-test measured using VAS, NDI, CCFT. Both the group received a hot pack for 10min as a common intervention.

On comparing the mean value of Group A & Group B on VAS and NDI Group B (neck stability with core stability exercise) showed 3.5 and 33.4 post-test values which were more effective than Group A (neck stability exercise) 5. 3 and 45.2 at P≤ 0.001. On the Craniocervical flexion Group B had shown 29.5 greater mean value when compared to Group A 24.7 at P≥ 0.001.

Higher proportions of patients improved in group B compared to group A. Core stability exercise group demonstrated and benefited significant improvements in NDI, VAS, and CCFT scores.

Mohsen et al., (2019) showed that 12 sessions of neck, core, and combined stabilization training in the neck region could improve the tolerance and pain of the elderly with non-specific chronic neck pain.

This is the first study to investigate the effect of adding IASTM to core stability exercise in treatment of mechanical neck pain.

Delimitation

This study was delimited to:

1. Subjects were divided randomly into two groups.
2. Age of the subjects ranged from 18 and 55 with mechanical neck pain.
3. Subjects were selected from outpatient clinic of Ismailia Medical Complex.
4. Pain level was measured by VAS.
5. Cervical range of motion and proprioception were measured using CROM.
6. Functions were measured by Arabic version of Neck Disability Index.
7. Muscle activity and H-reflex were measured by EMG. Basic Assumption

It was assumed that:

1. All subjects would exert their best effort to be relaxed during testing procedures.
2. All subjects would follow the researcher's instructions and advices.
3. Psychological condition would be the same for all subjects.

Hypotheses:

1. There would be no statistically significant effect of adding IASTM to core stability on pain level.
2. There would be no statistically significant effect of adding IASTM to core stability on cervical ROM.
3. There would be no statistically significant effect of adding IASTM to core stability on proprioception.
4. There would be no statistically significant effect of adding IASTM to core stability on muscle activity.
5. There would be no statistically significant effect of adding IASTM to core stability on H-reflex.
6. There would be no statistically significant effect of adding IASTM to core stability on functions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as having chronic mechanical neck pain.
2. Patient's age between 18-55 years old.

Exclusion Criteria:

1. Subjects with any specific neck pathology as radiculopathy, rheumatoid arthritis and systemic diseases.
2. sensory problems at mid or upper back.
3. A history of head and upper trunk trauma or surgery.
4. severe disorders of the cervical spine such as disk prolapse and cervical stenosis.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Pain level | 4 weeks
  The pain level was measured by visual analogue scale.The VAS is a 100-mm horizontal line anchored by word descriptors at each end by ''no pain'' on the left and ''worst imaginable pain'' on the right. The minimum score means it is better.
Cervical range of motion and proprioception | 4 weeks
  Cervical range of motion and proprioception were measured using CROM.
Functions | 4 weeks
  Functions were measured by Arabic version of Neck Disability Index. It is consisting of 10 items with six choices (0-5), Each item is scored from zero (no disability) to five (total disability). Minimum score means it is better.
Muscle activity | 4 weeks
  Muscle activity was measured by electromyography (EMG).
H-reflex | 4 weeks
  H-reflex was measured by EMG.

CONTACTS AND LOCATIONS:
Overall Officials: Haytham El-Hafez, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Ismailia Medical Complex, Ismailia, Egypt